CLINICAL TRIAL: NCT03083990
Title: Compare IBI305 to Avastin on the Pharmacokinetics, Safety, Tolerance and Immunogenicity of a Single Dose In Healthy Male Subjects: a Randomized Double-blind Parallel Controlled Phase I Clinical Study
Brief Title: Compare IBI305 and Bevacizumab on Pharmacokinetics/Safety/Immunogenicity on Healthy Male
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI305A201
Record Dates: First submitted 2016-11-12; First posted 2017-03-20 (Actual); Results first posted 2020-11-04 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Healthy
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): IBI 305 ,3mg/kg, infusion in 90 minutes
  Interventions: Biological: IBI305(Bevacizumab Biosimilar)
- Group B (Active Comparator): Bevacizumab (Avastin) 3mg/kg, infusion in 90 minutes
  Interventions: Drug: Avastin(Bevacizumab)

INTERVENTIONS:
Biological: IBI305(Bevacizumab Biosimilar) — 3mg/kg, infusion in 90minutes
  Arms: Group A
Drug: Avastin(Bevacizumab) — 3mg/kg, infusion in 90minutes
  Other Names: avastin
  Arms: Group B

SUMMARY:
To confirm the PK similarity of IBI305 and bevacizumab in healthy volunteers .

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for the study, patients should fulfill all the following criteria:

  1. Fully understand the study purpose, and understand the pharmacological effects and potential adverse reactions of the drug, voluntarily signed written informed consent according to the declaration of Helsinki.
  2. Age ≥18 and ≤ 50, healthy male subjects
  3. Weigh ≥ 50 kg and ≤ 100 kg， BMI≥ 19 and ≤ 28 kg/m2
  4. All the system test result within the normal range, or abnormal test results without clinical significance judged by the investigator.
  5. The subjects must agree to use effective contraceptive measures during the study treatment and for 6 months after receiving last does of study drug (e.g. abstinence, sterilization surgery, oral contraceptives, contraception by progesterone injection or subcutaneous)

Exclusion Criteria:

* Patients should not enter the study if any of the following exclusion criteria are fulfilled:

  1. Medical history of high blood pressure or abnormal blood pressure at screening/baseline(Double confirmed systolic blood pressure (SBP) >140 mmHg and/or diastolic blood pressure (DBP) > 90 mmHg within one day)
  2. Proteinuria with clinical significance judged by the investigator (routine urine examination, urine protein 2 + and above) or a history of proteinuria.
  3. Any prior VEGF(vascular endothelial growth factor) and VEGFR(Vascular Endothelial Growth Factor Receptor) antibody or protein treatment within one year.
  4. Any biological products or a live virus vaccine treatment within 3 months , or any monoclonal antibodies within 12 months before the first dose of study drug.
  5. History or evidence of inherited bleeding diathesis or coagulopathy or thrombus.
  6. History of digestive tract perforation or digestive tract fistula.
  7. Serious, non-healing wound, active ulcer, or untreated bone fracture, or major surgical procedure within 2 months prior to randomization or anticipation of need for major surgery during the course of the study or 2 months after last dose of the study drug.
  8. Use Rx or OTC drugs or nutritional health products within 5 half-lives or within 2 weeks before the first dose of study drug (According to the longer time).Herbal supplements need to stop at 28 days before the first dose of study drug.
  9. Positive hepatitis b surface antigen (HBsAg), hepatitis c virus (HCV) antibody, or human immunodeficiency virus (HIV) antibody or syphilis
  10. Known hypersensitivity to Bevacizumab or any excipients
  11. Known allergic disease or allergic constitution
  12. History of blood donation within 3 months before the first dose of study drug
  13. Treatment with any other investigational agent or participation in another clinical trial within 3 months prior to screening
  14. History of alcoholism or drug abuse within 12 months prior to screening; Subjects cannot temperance within 72 hours before study drug infusion and during the whole study
  15. History of mental illness
  16. Anticipated of partner pregnancy during the study.
  17. Incompliance to the clinical study protocol during the study.
  18. Other conditions that the investigator thinks unsuitable in this study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2017-08-17 (Actual); Study Completion 2017-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: yanhua Ding, Doctor, Principal Investigator — Jilin University First Hospital
Locations (1):
- Jilin University First Hospital, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- IBI305: IBI 305 ,3mg/kg, infusion in 90 minutes
  IBI305(Bevacizumab Biosimilar): 3mg/kg, infusion in 90minutes
- Bevacizumab: Bevacizumab (Avastin) 3mg/kg, infusion in 90 minutes
  Avastin(Bevacizumab): 3mg/kg, infusion in 90minutes
Period: Overall Study
Arm/Group | IBI305 | Bevacizumab
Started | 50 | 50
Completed | 49 | 50
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline demographics of the subjects were analyzed based on the Pharmacokinetics analysis set.A total of 98 (98.0%) subjects were included , and 2 (4%) subjects in the IBI305 arm were excluded in the due to positive anti-drug antibody at baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | IBI305 | Bevacizumab | Total
Number analyzed (Participants) | 48 | 50 | 98
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mean (SD) | 36.5 (8.92) | 34.0 (8.87) | 35.2 (8.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 48 | 50 | 98
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han | 43 | 45 | 88
  Others | 5 | 5 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  China | 48 | 50 | 98
Height [Mean (Standard Deviation); unit: centimeter] | 169.7 (5.69) | 169.0 (5.12) | 169.3 (5.39)
Weight [Mean (Standard Deviation); unit: kilogram] | 67.32 (7.763) | 68.42 (6.629) | 67.88 (7.191)
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 23.414 (2.739) | 23.962 (2.040) | 23.694 (2.412)

OUTCOME MEASURES:

1. Primary Outcome: AUC0 - t
Description: the area under the blood drug concentration time curve form 0 to t (AUC0 - t)
Time Frame: 60 min before intravenous infusion, 5 min after iv. infusion, 4 hr, 12 hr, 2 days, 3 days, 5 days, 8 days, 15 days, 22 days, 29 days, 43 days, 57 days, 64 days, 71 days, 85 days
Population: 2 subjects in the IBI305 arm were not included in the PKAS(PK analysis set) because of positive ADA at baseline
Measure: Geometric Mean (Standard Deviation); unit: h*ug/mL
Arm/Group | IBI305 | Bevacizumab
Number analyzed (Participants) | 48 | 50
h*ug/mL | 19704.2 (18.8) | 20736.9 (19.1)
Statistical Analysis 1: Comparison: IBI305 vs Bevacizumab; Test type: Equivalence — Geometric mean ratio and its 90%CI are obtained after anti-logarithmic transformation.If 90% CI for the geometric mean ratio of AUC 0-t and AUC 0-∞ (trial/control) ranges between 0.8-1.25, then it is considered that IBI305 and Bevacizumab are bioequivalent; p > 0.05, ANOVA; Odds Ratio (OR) = 0.9502, 90% CI 2-sided [0.8921 to 1.0120]

2. Primary Outcome: AUC0 - ∞
Description: the area under the blood drug concentration time curve form 0 to ∞AUC0 - ∞)
Time Frame: as for outcome 1
Population: 2 subjects in the IBI305 arm were not included in the PKAS(PK analysis set) because of positive ADA at baseline
Measure: Geometric Mean (Standard Deviation); unit: h*ug/mL
Arm/Group | IBI305 | Bevacizumab
Number analyzed (Participants) | 48 | 50
h*ug/mL | 20180.2 (18.6) | 21281.4 (19.8)
Statistical Analysis 1: Comparison: IBI305 vs Bevacizumab; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA; Odds Ratio (OR) = 0.9483, 90% CI 2-sided [0.8896 to 1.0108]

3. Secondary Outcome: Cmax
Description: Maximum serum concentration
Time Frame: as for outcome 1
Population: 2 subjects in the IBI305 arm were not included in the PKAS(PK analysis set) because of positive ADA at baseline
Measure: Geometric Mean (Standard Deviation); unit: ug/mL
Arm/Group | IBI305 | Bevacizumab
Number analyzed (Participants) | 48 | 50
ug/mL | 65.3 (21.0) | 67.0 (18.9)
Statistical Analysis 1: Comparison: IBI305 vs Bevacizumab; Test type: Equivalence; p > 0.05, ANOVA; Odds Ratio (OR) = 0.9749, 90% CI 2-sided [0.9123 to 1.0418]

4. Secondary Outcome: t1/2
Description: elimination half life
Time Frame: as for outcome 1
Population: 2 subjects in the IBI305 arm were not included in the PKAS(PK analysis set) because of positive ADA at baseline
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | IBI305 | Bevacizumab
Number analyzed (Participants) | 48 | 50
hour | 340.2 (51.1) | 356.5 (69.6)

5. Secondary Outcome: Clearance Rate
Description: apparent clearance
Time Frame: as for outcome 1
Population: 2 subjects in the IBI305 arm were not included in the PKAS(PK analysis set) because of positive ADA at baseline
Measure: Mean (Standard Deviation); unit: ml/h/kg
Arm/Group | IBI305 | Bevacizumab
Number analyzed (Participants) | 48 | 50
ml/h/kg | 0.151 (0.0296) | 0.144 (0.0281)

6. Secondary Outcome: Apparent Volume of Distribution
Description: apparent volume of distribution(V）
Time Frame: as for outcome 1
Population: 2 subjects in the IBI305 arm were not included in the PKAS(PK analysis set) because of positive ADA at baseline
Measure: Mean (Standard Deviation); unit: ml/kg
Arm/Group | IBI305 | Bevacizumab
Number analyzed (Participants) | 48 | 50
ml/kg | 73.8 (15.9) | 72.3 (12.8)

7. Other Pre Specified Outcome: Number of Participants Positive for Nab（Neutralizing Antibody）
Description: The analysis of NAb was done by Covance Pharmaceutical R&D (Shanghai) Co., Ltd. using methodologically validated ECL immunoassay.
Time Frame: 99 days after administration
Population: All 100 (100%) subjects were included in the NAb-AS (Neutralizing anti-body analysis set)
Measure: Number; unit: Participants
Arm/Group | IBI305 | Bevacizumab
Number analyzed (Participants) | 50 | 50
Participants
  Baseline | 2 | 0
  D15 | 4 | 0
  D43 | 2 | 0
  D71 | 2 | 0
  D99 | 1 | 0

8. Other Pre Specified Outcome: Number of Participants Positive for Anti-drug Antibodies
Description: The analysis of ADA was done by Wuxi AppTec (Shanghai) Co., Ltd. using methodologically validated electrochemiluminescence (ECL) immunoassay.
Time Frame: 99 days after administration
Population: All 100 (100%) subjects were included in the ADA-AS(Anti-drug Antibody Analysis set)
Measure: Number; unit: Participants
Arm/Group | IBI305 | Bevacizumab
Number analyzed (Participants) | 50 | 50
Participants
  Baseline | 2 | 0
  D15 | 4 | 0
  D43 | 2 | 0
  D71 | 2 | 0
  D99 | 1 | 0

9. Other Pre Specified Outcome: Systolic Blood Pressure
Description: Systolic blood pressure and diastolic blood pressure on certain timepoints are measured and recorded.
Time Frame: 0, D1( immediately after the end of infusion), D1 (4 hrs after the start of infusion), D1, 8 hrs after the start of infusion, D1 (12 hrs after the start of infusion), D2, D3, D5, D8, D15, D22, D29, D43, D57, D64, D71, D85, D99
Population: All 100 (100%) subjects were included in the safety analysis set. Blood pressure of certain timepoint was not collected because of serve adverse event.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | IBI305 | Bevacizumab
Number analyzed (Participants) | 50 | 50
mmHg
  Baseline | 119.6 (8.73) | 121.4 (8.02)
  D1, immediately after the end of infusion | 113.3 (10.23) | 114.5 (8.7)
  D1, 4 hrs after the start of infusion | 118.0 (9.60) | 119.6 (7.87)
  D1, 8 hrs after the start of infusion | 120.4 (9.48) | 120.3 (8.30)
  D1, 12 hrs after the start of infusion | 119.8 (8.67) | 123.4 (9.63)
  D2 | 119.8 (9.72) | 121.9 (8.81)
  D3 | 120.2 (8.37) | 123.2 (9.52)
  D5 | 120.7 (7.97) | 121.4 (8.34)
  D8 | 118.4 (7.69) | 122.6 (9.22)
  D15 | 118.6 (9.70) | 118.5 (10.19)
  D22 | 121.8 (8.73) | 122.5 (8.88)
  D29 | 121.6 (9.20) | 123.1 (8.91)
  D43 | 119.7 (9.12) | 121.3 (9.03)
  D57 | 118.4 (10.30) | 122.1 (8.12)
  D64: number analyzed (Participants) | 49 | 50
  D64 | 119.4 (8.78) | 120.2 (10.00)
  D71: number analyzed (Participants) | 49 | 50
  D71 | 118.3 (10.01) | 119.8 (10.10)
  D85: number analyzed (Participants) | 49 | 50
  D85 | 115.8 (9.04) | 120.6 (9.59)
  D99: number analyzed (Participants) | 49 | 50
  D99 | 118.2 (7.61) | 118.2 (10.66)

10. Other Pre Specified Outcome: Diastolic Blood Pressure
Description: Systolic blood pressure and diastolic blood pressure on certain timepoints are measured and recorded.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | IBI305 | Bevacizumab
Number analyzed (Participants) | 50 | 50
mmHg
  Baseline | 79.2 (8.02) | 81.4 (5.94)
  D1, immediately after the end of infusion | 71.8 (7.82) | 73.7 (6.64)
  D1, 4 hrs after the start of infusion | 75.5 (6.68) | 77.4 (7.13)
  D1, 8 hrs after the start of infusion | 77.8 (5.94) | 79.3 (6.95)
  D1, 12 hrs after the start of infusion | 77.0 (6.96) | 81.3 (7.37)
  D2 | 79.8 (6.57) | 81.6 (6.46)
  D3 | 80.5 (6.45) | 82.8 (6.17)
  D5 | 80.4 (8.30) | 82.1 (4.71)
  D8: number analyzed (Participants) | 50 | 49
  D8 | 78.2 (6.23) | 81.4 (6.62)
  D15 | 78.2 (7.67) | 79.2 (6.50)
  D22 | 80.5 (6.04) | 82.3 (7.47)
  D29 | 79.6 (6.43) | 81.6 (7.02)
  D43 | 79.5 (7.34) | 80.0 (6.96)
  D57 | 78.6 (7.87) | 82.2 (6.18)
  D64: number analyzed (Participants) | 49 | 50
  D64 | 78.7 (7.33) | 80.5 (6.18)
  D71: number analyzed (Participants) | 49 | 50
  D71 | 77.1 (8.01) | 80.2 (6.32)
  D85: number analyzed (Participants) | 49 | 50
  D85 | 79.2 (6.96) | 80.0 (6.42)
  D99: number analyzed (Participants) | 49 | 50
  D99 | 76.8 (6.91) | 77.9 (6.83)

11. Other Pre Specified Outcome: Urinalysis
Description: Urine specific gravity as assessed by laboratory tests up to 99 days post-treatment
Time Frame: Baseline,D2,D5,D15,D29,D57,D71,D99
Population: All 100 (100%) subjects were included in the analysis set
Measure: Mean (Standard Deviation); unit: Urine specific gravity
Arm/Group | IBI305 | Bevacizumab
Number analyzed (Participants) | 50 | 50
Urine specific gravity
  Baseline | 1.017 (0.006) | 1.017 (0.006)
  D2 | 1.017 (0.006) | 1.017 (0.005)
  D5 | 1.017 (0.005) | 1.018 (0.005)
  D15 | 1.016 (0.006) | 1.017 (0.006)
  D29 | 1.017 (0.005) | 1.017 (0.005)
  D57 | 1.016 (0.005) | 1.018 (0.006)
  D71 | 1.017 (0.004) | 1.016 (0.005)
  D99 | 1.017 (0.006) | 1.019 (0.006)

12. Other Pre Specified Outcome: Hemoglobin
Description: Hemoglobin as assessed by laboratory tests up to 99 days post-treatment.
Time Frame: Baseline,D2,D5,D15,D29,D57,D71,D99
Population: All 100 (100%) subjects were included in the safety analysis set (SS)
Measure: Mean (Standard Deviation); unit: Hemoglobin (g/L)
Arm/Group | IBI305 | Bevacizumab
Number analyzed (Participants) | 50 | 50
Hemoglobin (g/L)
  Baseline | 161.0 (9.42) | 163.5 (9.52)
  D2 | 158.8 (11.53) | 160.4 (9.21)
  D5 | 165.4 (10.93) | 167.7 (10.02)
  D15 | 160.9 (10.67) | 164.5 (9.21)
  D29 | 161.1 (10.01) | 164.5 (11.03)
  D57 | 160.4 (12.45) | 165.5 (10.42)
  D71 | 159.8 (12.19) | 163.9 (9.12)
  D99 | 154.6 (11.01) | 159.9 (10.22)

ADVERSE EVENTS:
Time Frame: from participants are enrolled to 99 days after infusion
Description: The analysis population consisted of all participants.
Arm/Group | IBI305 | Bevacizumab
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/50 | 0/50
Other Adverse Events (participants affected / at risk) | 40/50 | 40/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IBI305 (N=50) | Bevacizumab (N=50)
hand injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IBI305 (N=50) | Bevacizumab (N=50)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 11 (25) | 13 (24)
ALT increased (Investigations) | 10 (12) | 12 (17)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (8) | 9 (11)
AST increased (Investigations) | 6 (8) | 10 (12)
White blood cell count increased (Investigations) | 6 (9) | 8 (9)
Neutrophil count increased (Investigations) | 5 (7) | 8 (9)
Sinus bradycardia (Cardiac disorders) | 4 (6) | 3 (4)
White blood cell count decreased (Investigations) | 4 (7) | 2 (5)
Red blood cells urine positive (Investigations) | 4 (4) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (5) | 3 (8)
Headache (Nervous system disorders) | 3 (4) | 0 (0)
Intermediate insomnia (Psychiatric disorders) | 3 (3) | 0 (0)
Bilirubin increased (Investigations) | 2 (3) | 6 (8)
White blood cells urine positive (Investigations) | 2 (3) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-08-03): https://cdn.clinicaltrials.gov/large-docs/90/NCT03083990/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT03083990/SAP_001.pdf